CLINICAL TRIAL: NCT00441376
Title: A Phase I Dose Escalation Tolerability Study of ThermoDox™ (Thermally Sensitive Liposomal Doxorubicin) in Combination With Radiofrequency Ablation (RFA) of Primary and Metastatic Tumors of the Liver
Brief Title: A Study of ThermoDox™ in Combination With Radiofrequency Ablation (RFA) in Primary and Metastatic Tumors of the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imunon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-06-101-01
Record Dates: First submitted 2007-02-26; First posted 2007-02-28 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma; Liver Neoplasms
Keywords: Radiofrequency ablation; RFA; Doxorubicin; Liposome; HCC; MLC; hepatocellular carcinoma; liver tumor; tumor; ablation; heat therapy; anti-tumor; liver cancer; metastatic liver cancer (MLC)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms; Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ThermoDox + RFA (Experimental): ThermoDox administered as single dose intravenously over 30 minutes in combination with radiofrequency ablation. Dose is determined by dose cohort patient enters study.
  Interventions: Drug: ThermoDox

INTERVENTIONS:
Drug: ThermoDox — 15 ml vial containing 2mg/ml Doxorubicin HCl, DPPC, MSPC, DSPE-MPEG 2000. Administered as single dose intravenously over 30 minutes. Dose is determined by dose cohort patient enters study.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) of ThermoDox when used in combination with radiofrequency ablation (RFA) in the treatment of primary and metastatic tumors of the liver.

DETAILED DESCRIPTION:
Ablative treatment approaches, such as RFA or microwave ablation, have received increased attention as alternates to other treatment approaches such as hepatic arterial embolization or chemoembolization (TACE) or percutaneous ethanol injection (PEI) in the majority of patients who are either not candidates for surgical resection or are not offered palliative supportive care only for diffuse disease. RFA can be applied repetitively to the same patient to treat multiple tumors at time of diagnosis or upon tumor recurrence (local or distant to the site of ablation), and is largely limited in its application only by tumor location and size (tumors near larger vessels, bowel or the hepatobiliary tree are more difficult to ablate). To extend the volume of the ablation region in a controlled fashion in patients and to improve the ability to kill tumor cells in the ablation margin region and allow for the improved treatment of HCC and MLC lesions > 3 cm in diameter by complete thermal ablation, Celsion Corporation has developed ThermoDox, a thermally sensitive, intravenously administered liposomal formulation of doxorubicin capable of selectively releasing its drug contents when exposed to temperatures of > 39.5°C. The concept behind this treatment approach is to create a large concentration gradient of doxorubicin in the immediate region of the tumor which borders the zone of RFA induced cell necrosis. The temperature isotherms produced in this boundary region should be adequate to activate doxorubicin release by the thermally sensitive liposomes deposited locally around the ablation zone. This in effect increases the region of tissue that can be treated beyond that achievable by RFA alone. Several clinical objectives are being tested in this study. The MTD for ThermoDox is to be confirmed. This study will assess the safety of using ThermoDox in conjunction with RFA over multiple cycles, consistent with the clinical needs of the subjects. While this study is not powered to define effectiveness of the combination of RFA plus ThermoDox, the results of this study should allow for an assessment of risk and benefit for designing future studies. This study will also test alternative infusion reaction prophylaxis regimens.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Are willing to sign an informed consent form, indicating that they are aware of the investigational nature of this study that is in keeping with the policies of the institution.
* Have a diagnosis of metastatic liver cancer (MLC) or primary hepatocellular cancer (HCC) confined to the liver.
* Be an appropriate candidate for receiving RFA as a medically indicated treatment.
* Have an echocardiogram revealing an Ejection Fraction (EF) ≥ 50%.
* Willing to return to the study site for their imaging scans.
* Have life expectancy of ≥ 3 months.
* Have ECOG performance status of 0-2 or Karnofsky score of 60-100% (see Appendix II).
* Have no more than Childs-Pugh Class B liver disease.
* Subjects must have no prior doxorubicin exposure.
* No single lesion should be > 7 cm in maximum diameter.
* Subjects must agree to receive no other systemic therapy from the time of study enrollment until a minimum of 21 days after their ThermoDox infusion

Exclusion Criteria:

* Have serious medical illnesses including, but not limited to, congestive heart failure, myocardial infarction or cerebral vascular accident within the last six months, or life threatening cardiac arrhythmias.
* Are pregnant or breast feeding. In women of childbearing potential, a negative pregnancy test (serum) is required at baseline, 1 month and each 3 month follow-up visit.
* Are not practicing an acceptable form of birth control (i.e. diaphragm, cervical cap, condom, surgical sterility or birth control pills. Woman whose husband has undergone a vasectomy must use a second form of birth control).
* Have known serious allergic reactions (anaphylaxis) to any of the drugs or liposomal components or imaging agents to be used in this study.
* Have portal or hepatic vein invasion/thrombosis.
* Have PT or PTT > 1.5 times the institution's upper normal limit (UNL), except in subjects who are therapeutically anticoagulated for non-related medical conditions such as atrial fibrillation.
* Have platelet count > 75,000/mm3, absolute neutrophil count > 1500/mm3, or Hgb > 10 (unless the hemoglobin value has been stable, the subject is cardiovascularly stable, asymptomatic and judged able to withstand the RFA
* Have serum creatinine ≤ 2.0 mg/dl (or calculated CrCl ≤ 60mL/min).
* Have contraindications to receiving doxorubicin HCl.
* Are being treated with other investigational agents (within a minimum of 30 days or 5 half-lives of the investigational agent).
* Have other concurrent malignancy (subjects with benign or non aggressive malignant tumors-e.g.: squamous cell cancer of the skin-may be included), evidence of extrahepatic cancer from their primary malignancy, or ongoing, medically significant active infection.
* Documented HIV positive.
* NYHA class III or IV cardiovascular disease or LVEF < 50%.
* Evidence of hemachromatosis.
* Are on any of the medications listed in section 6.3, which could have an adverse effect when combined with the study drug, and who cannot stop the medication for the duration of the study and 30 days beyond the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of systemically delivered, heat-activated liposome encapsulated doxorubicin (ThermoDox) in combination with radiofrequency ablation (RFA) of liver neoplasms. | 1 month
To test alternative infusion reaction prophylaxis regimens | 48 hours
To assess the safety of ThermoDox plus RFA afer administration of potential multiple cycles | 3 years
To determine the Pharmacokinetics (PK) of ThermoDox | 48 hours

SECONDARY OUTCOMES:
To document any anti-tumor activity and assess recurrences. | 3 years
To measure post ablation lesion volume. | 1 month
To determine the cardiotoxicity of ThermoDox through enhanced ECG monitoring. | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Northshore Hospital - Long Island Jewish Health System, Manhasset, New York, United States